CLINICAL TRIAL: NCT01922219
Title: Predictors of Treatment Outcome With Cognitive Behavioral Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6127; 5K08MH085061 (NIH)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorder
Keywords: depression; cognitive therapy; cognitive behavioral therapy; CBT; psychotherapy; MDD; major depressive disorder; MRI; fMRI
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Behavioral Therapy (Other): Depressed individuals who enroll in this study will receive 14 sessions of cognitive behavioral therapy provided by an experienced psychiatrist or psychologist over 12 weeks (twice-a-week for the first two weeks, and weekly after that).
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 14 sessions of individual psychotherapy (cognitive behavioral therapy) for depression over 12 weeks

SUMMARY:
The purpose of this research study is to learn whether specific types of brain imaging and psychological testing can predict how much benefit patients with depression will receive from a well-studied psychotherapy for depression, called cognitive behavioral therapy (CBT), and how the brain imaging and psychological tests change with treatment. We will also be comparing brain scans from this study between individuals suffering from depression and volunteers without depression.

This study offers 14 sessions of one-on-one cognitive-behavioral therapy (CBT) over twelve weeks, administered by an experienced doctoral-level psychologist or psychiatrist.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) affects 13.1 - 14.2 million American adults annually. Cognitive-behavioral therapy (CBT) is a structured psychotherapy that has been demonstrated in multiple studies to be an effective treatment for MDD. Not all patients achieve a full remission from MDD with CBT, however. Mental health clinicians currently lack clinical or biological markers that can reliably predict treatment outcome with CBT for MDD. Developing such markers could greatly improve clinical outcomes, and could facilitate matching of patients to treatments that are likely to help them. A recent functional magnetic resonance imaging (fMRI) study in healthy individuals examined the neural correlates of cognitive strategies to regulate emotional responses to emotional stimuli. The emotional regulation techniques used in this fMRI study map closely onto the cognitive restructuring techniques that are a primary tool used in CBT for MDD. There is evidence that patients with depression may benefit most from a psychotherapy that draws on their existing strengths. We therefore propose to examine the neural representations of emotion regulation as a predictor of treatment outcome with CBT for MDD. We will recruit subjects with MDD in a current major depressive episode. Research participants will complete baseline psychological and biological assessments, including MRI and functional MRI imaging. Following scanning, subjects will receive 14 sessions of individual CBT for depression over 12 weeks, administered by an experienced psychiatrist or psychologist. Baseline assessments will be examined as predictors of treatment outcome with CBT for depression.

ELIGIBILITY:
Inclusion Criteria:

* In a current major depressive episode
* If currently on medications, lack of benefit after an adequate trial. If currently on medications, willing and able to tolerate a medication washout.
* Ability to provide an informed consent
* For healthy volunteers, no current or past history of depression

Exclusion Criteria:

* Unstable medical conditions
* Current alcohol or substance abuse or dependence
* Current or past history of other major psychiatric disorders such as Bipolar disorder, schizophrenia, or other psychotic illnesses (Anxiety in depressed participants is okay)
* For females, current pregnancy
* Dementia or neurological disease or head trauma with evidence of cognitive impairment
* Currently taking fluoxetine
* Contraindication to CBT
* Presence of metal in body
* Claustrophobia
* Weight > 350 pounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Miller, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pantazatos SP, Yttredahl A, Rubin-Falcone H, Kishon R, Oquendo MA, John Mann J, Miller JM. Depression-related anterior cingulate prefrontal resting state connectivity normalizes following cognitive behavioral therapy. Eur Psychiatry. 2020 Apr 14;63(1):e37. doi: 10.1192/j.eurpsy.2020.34. PMID 32284075

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy
Started | 37
Completed | 28
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Cognitive Behavioral Therapy
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 3
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Remitters as Assessed by Post-treatment Beck Depression Inventory Less Than or Equal to 10
Description: The primary outcome of this study is remission from depression at the conclusion of 12 weeks of cognitive behavioral therapy for depression. This will be assessed using the Beck Depression Inventory, a self-report questionnaire of symptoms of depression that will be administered at every treatment visit. Remission is defined by a final Beck Depression Inventory score less than or equal to 10.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioral Therapy
Number analyzed (Participants) | 37
Participants | 13

2. Secondary Outcome: Post-Treatment Beck Depression Inventory
Description: The Beck Depression Inventory is a self-report measure of depression severity that is a well-characterized scale with excellent psychometric properties and is frequently used in research studies of depression.
  The scale measures symptoms related to sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, changes in sleeping pattern, irritability, changes in appetite, concentration difficulty, tiredness or fatigue, and loss of interest in sex.
  We report the total score on the BDI, which has a range of 0 to 63. Higher values represent greater severity of depression. The following score interpretations are provided in the scale's manual:
  0-9 minimal depression 10-18 mild depression 19-29 moderate depression 30-63 severe depression
Time Frame: Post-Treatment, up to 12 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cognitive Behavioral Therapy
Number analyzed (Participants) | 37
Score on a scale | 15.4 (9.5)

3. Secondary Outcome: Final Score on the Hamilton Depression Rating Scale
Description: Final score on the Hamilton Depression Rating Scale (HDRS) was calculated for 37 patients who were treated with Cognitive Behavioral Therapy.
  The 17-item HDRS is a clinician-administered scale that quantifies depression severity, and includes items assessing mood, suicidal thinking, insomnia, feelings of guilt, work and activities, somatic symptoms, and insight. It is a well-characterized scale with excellent psychometric properties. The total score is the sum of the individual scores of the 17 scale items. Higher scores indicate greater depression severity. When using this outcome measure, we covary for baseline HDRS scores. Published norms for interpretation of the 17-item HDRS use a different version of the scale with a total possible score of 52, and are listed below. Interpretation is comparable (but not identical) with the 17-item HDRS version used in this study, which has a maximum score is 51.
  None: 0-7 Mild: 8-13 Moderate: 14-19 Severe: 20-25 Very Severe: 26-52
Time Frame: Post-Treatment, up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy
Number analyzed (Participants) | 37
units on a scale | 13.41 (6.61)

ADVERSE EVENTS:
Arm/Group | Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 1/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (N=37)
Knee Pain during MRI (Injury, poisoning and procedural complications) | 1 (1) — During an MRI, a subject developed mild unilateral knee pain similar to pain she had experienced in the past, and subsequently developed some stiffness and swelling in this knee. The IRB concluded that the event was neither serious nor study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes